CLINICAL TRIAL: NCT07128017
Title: Efficacy and Mechanisms of Internet-delivered MBCT for Adjustment Disorder During the COVID-19 Pandemic: A Randomized Controlled Trial
Brief Title: Online MBCT for Adjustment Disorder During COVID-19: Efficacy, Mechanisms, and RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warsaw (Other)
Responsible Party: Principal Investigator, Paweł Holas, MD, PhD, University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UWarsaw1
Record Dates: First submitted 2025-08-15; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Adjustment Disorder; Anxiety; Depressive
Keywords: Adjustment Disorder; Mindfulness-Based Cognitive Therapy; MBCT; Internet-delivered intervention; Online mental health; Cognitive defusion; Self-compassion; Experiential avoidance; Progressive Muscle Relaxatio; COVID-19 pandemic; Stress-related disorders; Depression; Anxiety; Randomized controlled trial; Unguided self-help interventio
MeSH Terms: conditions — Adjustment Disorders; Anxiety Disorders; COVID-19; Depression | interventions — Mindfulness-Based Cognitive Therapy; Autogenic Training

STUDY DESIGN:
Intervention Model Description: his study used a three-arm, parallel-group randomized controlled trial design. Participants meeting ICD-11 criteria for Adjustment Disorder were randomly assigned to one of three conditions: (1) unguided internet-delivered Mindfulness-Based Cognitive Therapy (iMBCT), (2) internet-delivered Progressive Muscle Relaxation (iPMR) as an active control, or (3) a waitlist control (WLC). Randomization was stratified by demographic characteristics and baseline symptom severity to ensure balanced groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet-Delivered Mindfulness-Based Cognitive Therapy (iMBCT) (Experimental): Internet-Delivered Mindfulness-Based Cognitive Therapy (iMBCT) Participants received a 4-week, unguided online adaptation of Mindfulness-Based Cognitive Therapy. The program consisted of six sequential modules delivered via a secure web platform, introducing mindfulness meditation, body scan, mindful movement, and cognitive-behavioral exercises. Content was provided through audio recordings, written materials, and reflective exercises. Supportive reminder emails were sent, but no therapist guidance was given.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (Internet-delivered)
- Internet-Delivered Progressive Muscle Relaxation (iPMR) (Active Comparator): Participants received a 4-week, unguided online progressive muscle relaxation program adapted from Bernstein and Borkovec's protocol. The program consisted of six sequential modules teaching systematic tensing and releasing of major muscle groups, gradually reducing the number of groups over time until relaxation could be achieved through recall alone. Audio guidance, written instructions, and reminder emails were provided without therapist involvement.
  Interventions: Behavioral: Progressive Muscle Relaxation (Internet-delivered)
- Waitlist Control (WLC) (Placebo Comparator): Participants were placed on a 4-week waitlist without active intervention. They completed all study assessments on the same schedule as intervention arms. At the end of the waiting period, they were offered the choice to participate in either the iMBCT or iPMR program.
  Interventions: Behavioral: No Intervention - Waitlist Control

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy (Internet-delivered) — A 4-week (30 days), unguided online adaptation of the Mindfulness-Based Cognitive Therapy (MBCT) program. The intervention consisted of six sequential modules delivered through a secure web platform, including guided mindfulness meditations, body scan, mindful movement, and cognitive-behavioral exercises. Participants received audio recordings, written materials, and reflective tasks, along with automated reminder emails. No therapist guidance was provided.
  Other Names: iMBCT
  Arms: Internet-Delivered Mindfulness-Based Cognitive Therapy (iMBCT)
Behavioral: Progressive Muscle Relaxation (Internet-delivered) — A 4-week, unguided online progressive muscle relaxation (PMR) program adapted from Bernstein and Borkovec's protocol. The program included six sequential modules teaching systematic tensing and relaxing of major muscle groups, gradually reducing the number of groups until relaxation could be achieved through recall alone. Materials included audio recordings, written instructions, and automated reminder emails. No therapist guidance was provided.
  Other Names: iPMR
  Arms: Internet-Delivered Progressive Muscle Relaxation (iPMR)
Behavioral: No Intervention - Waitlist Control — Participants in this arm received no active intervention during the 4-week waitlist period but completed all study assessments on the same schedule as intervention arms. After the waiting period, participants were offered the choice to take part in either the online MBCT or PMR program.
  Arms: Waitlist Control (WLC)

SUMMARY:
This study tested a 4-week, internet-based Mindfulness-Based Cognitive Therapy (MBCT) program designed to help people experiencing adjustment disorder during the COVID-19 pandemic. Adjustment disorder is a stress-related condition that can cause anxiety, depression, and difficulty coping after major life changes.

We compared the online MBCT program to two other groups: an internet-based relaxation training program and a wait-list group. A total of 301 adults from Poland took part. We measured symptoms of adjustment disorder, depression, and anxiety before the program, right after, and one month later.

Results showed that the online MBCT program led to greater improvements in depression and anxiety than the other two groups. People in MBCT also developed more self-compassion and were better able to distance themselves from unhelpful thoughts, which helped reduce their symptoms. Benefits lasted at least one month after the program ended.

These findings suggest that a brief, self-guided, online mindfulness program can be an effective, accessible way to support mental health during stressful times such as a pandemic.

DETAILED DESCRIPTION:
Background and Rationale Adjustment disorder (AjD) is a stress-related mental health condition characterized by maladaptive emotional and behavioral responses to an identifiable stressor. Core symptoms include persistent preoccupation with the stressor and difficulty adapting, often accompanied by anxiety, depressed mood, and avoidance behaviors. According to ICD-11 criteria, AjD symptoms emerge within three months of a stressor and typically resolve within six months after the stressor ends, although in many cases they can persist longer and contribute to chronic distress.

Epidemiological studies indicate that AjD is highly prevalent, affecting up to 30% of clinical populations and a substantial proportion of the general public during times of widespread stress. Despite this, AjD remains understudied compared to mood and anxiety disorders. Few empirically validated psychological interventions are available, and existing treatment recommendations are often extrapolated from evidence on depression and anxiety.

The COVID-19 pandemic presented a unique context in which AjD rates surged globally. Fear of infection, prolonged social isolation, economic uncertainty, and disruption of daily life contributed to high levels of stress-related distress. Surveys during the pandemic indicated that 18-43% of adults in Europe reported symptom patterns consistent with AjD, underscoring the urgent need for scalable interventions that could be delivered remotely and at low cost.

Mindfulness-Based Cognitive Therapy (MBCT) MBCT is an eight-week, group-based psychological program originally developed to prevent relapse in recurrent depression. It combines mindfulness meditation practices with cognitive-behavioral therapy strategies, fostering non-judgmental awareness of present-moment experience, greater cognitive flexibility, and reduced reactivity to negative thoughts and emotions.

Mechanistic research suggests that MBCT works by:

Increasing cognitive defusion - the ability to step back from and observe thoughts without automatically believing or reacting to them.

Reducing experiential avoidance - the tendency to suppress or avoid difficult emotions and sensations.

Enhancing self-compassion - a kinder, more understanding stance toward oneself in times of suffering.

These processes are relevant to AjD, where stressor-related rumination and self-critical coping often maintain distress. Although MBCT's efficacy for depression and anxiety is well-established, little is known about its effects in AjD or its feasibility in brief, fully online, self-guided formats.

Internet-Delivered MBCT (iMBCT) Internet-delivered psychological interventions (IPIs) have the potential to greatly expand access to evidence-based care. Online MBCT (iMBCT) can be delivered synchronously (live sessions with a facilitator) or asynchronously (self-paced, unguided), with evidence supporting effectiveness in reducing distress and improving resilience. Unguided iMBCT programs are especially promising for public health implementation due to their low delivery cost and scalability, but high-quality trials in specific clinical groups remain rare.

Study Objectives

The primary aim of this study was to evaluate the efficacy of a four-week, unguided, internet-delivered MBCT program for adults meeting ICD-11 criteria for AjD during the COVID-19 pandemic. We compared iMBCT with:

An active control - a four-week, unguided internet-delivered Progressive Muscle Relaxation (iPMR) program.

A passive control - a wait-list control (WLC).

Secondary aims were to examine whether changes in key psychological processes (cognitive fusion, experiential avoidance, self-compassion) mediated symptom improvement, providing insight into the mechanisms through which iMBCT exerts its effects.

Methods Overview This was a three-arm, parallel-group randomized controlled trial. A total of 301 adults from Poland who met ICD-11 AjD criteria (based on the Adjustment Disorder New Module - 20) were randomized to iMBCT, iPMR, or WLC. Interventions lasted four weeks, with assessments at baseline, post-intervention, and one-month follow-up (for intervention groups).

Interventions

iMBCT: A self-guided adaptation of MBCT condensed to six modules over 30 days. Modules included audio-guided mindfulness meditations (body scan, sitting meditation, mindful movement), reflective journaling, and psychoeducational materials. Content was delivered through a secure online platform with automated email reminders.

iPMR: A self-guided Progressive Muscle Relaxation program based on the Bernstein and Borkovec protocol, progressing from tensing and releasing 16 muscle groups to relaxation through mental recall. Audio instructions and written materials were provided.

WLC: No intervention during the 4-week study period. Participants were offered a choice of iMBCT or iPMR afterward.

Outcomes and Process Measures

Primary outcomes:

AjD symptoms (ADNM-20)

Depressive symptoms (PHQ-9)

Anxiety symptoms (GAD-7)

Process measures:

Cognitive Fusion (CFQ)

Experiential Avoidance (AAQ-II)

Self-Compassion (SCS-SF)

Key Findings

All groups showed significant symptom reductions over time, but iMBCT participants had greater improvements in depression and anxiety than both iPMR and WLC.

AjD remission rates were highest in the iMBCT group.

Cognitive defusion fully mediated the effect of iMBCT on depression and anxiety, suggesting it is a key mechanism of change.

Increases in self-compassion were observed only in the iMBCT group compared to WLC.

Benefits in the intervention groups were maintained at one-month follow-up.

Significance and Implications This trial provides the first randomized evidence that a brief, unguided iMBCT program can effectively reduce symptoms of AjD, depression, and anxiety, and improve transdiagnostic processes associated with resilience. Its low cost, scalability, and sustained benefits make it a promising tool for addressing stress-related disorders in situations where traditional face-to-face therapy is unavailable or impractical, such as during large-scale public health crises.

The findings also add to the mechanistic literature on MBCT, highlighting cognitive defusion as a central pathway to symptom improvement in AjD. This may inform refinements in mindfulness-based interventions and encourage further research on tailoring MBCT to specific stressor-related conditions.

Future research should test longer-term outcomes, evaluate implementation in diverse cultural contexts, and explore the integration of brief guidance or peer support to reduce attrition.

ELIGIBILITY:
Inclusion Criteria:

Participants are required to be (a) at least 18 years old, (b) have access to the Internet, (c) currently experiencing some form of psychological distress related to COVID-19 pandemic, such as stress, anxiety, and/or low mood, and d) have the willingness to commit to a free online intervention program with two pre and post measurements online, within four weeks.

Exclusion Criteria:

(a) participating simultaneously in any pharmaceutical or psychosocial therapy, (b) if they were suffering from a current or lifetime psychotic disorder, bipolar disorder, or substance abuse problem; (c) if they reported current suicidal tendencies, (d) if they did not meet criteria for Adjustment Disorder (less than 47,5 points in ADNM-20 questionnaire), (e) participated in the past or currently in any of 8 weeks mindfulness programs (e.g., MBSR, MBCT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Change in Adjustment Disorder symptoms | Baseline (Week 0) and Post-intervention (Week 4)
  Change in Adjustment Disorder symptoms from baseline to post-intervention, measured by the Adjustment Disorder New Module - 20 (ADNM-20).
  The ADNM-20 is a validated self-report questionnaire assessing ICD-11 Adjustment Disorder symptoms, including preoccupation and failure to adapt. Scores range from 0 to 60, with higher scores indicating greater symptom severity.
Remission Rates from Adjustment Disorder | Baseline (Week 0) and Post-intervention (Week 4)
  Instrument: Adjustment Disorder New Module - 20 (ADNM-20) Proportion of participants scoring below the clinical cutoff (>47.5) on the ADNM-20 at post-intervention, indicating remission from probable Adjustment Disorder.

SECONDARY OUTCOMES:
Change in Depressive Symptoms | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 8)
  Patient Health Questionnaire-9 (PHQ-9). Description: The PHQ-9 is a validated self-report measure assessing the severity of depressive symptoms. Scores range from 0 to 27, with higher scores indicating greater severity.
Change in Anxiety Symptoms | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 8)
  Instrument: Generalized Anxiety Disorder Scale-7 (GAD-7) The GAD-7 is a validated self-report measure of generalized anxiety symptoms. Scores range from 0 to 21, with higher scores indicating greater severity.
Change in Cognitive Fusion | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 8)
  Instrument: Cognitive Fusion Questionnaire (CFQ). The CFQ assesses the extent to which individuals are entangled with their thoughts. Scores range from 7 to 49, with higher scores indicating greater cognitive fusion.
Change in Self-Compassion | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 8)
  Instrument: Self-Compassion Scale - Short Form (SCS-SF). Description: The SCS-SF measures self-compassion across six subdomains. Scores range from 12 to 60, with higher scores indicating greater self-compassion.
Change in Experiential Avoidance | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 8)
  Instrument: Acceptance and Action Questionnaire - II (AAQ-II). The AAQ-II measures experiential avoidance (the tendency to avoid unpleasant thoughts and feelings). Scores range from 7 to 49, with higher scores indicating greater avoidance.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology, University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
At this time, it has not been determined whether individual participant data (IPD) will be shared. The decision will depend on considerations such as participant privacy, applicable legal and ethical requirements, and the availability of resources to prepare de-identified datasets.